CLINICAL TRIAL: NCT01325480
Title: High Septal Pacing for Cardiac Resynchronization Therapy Acute Research Study
Brief Title: High Septal Pacing for Cardiac Resynchronization Therapy
Acronym: HISTORY
Status: Terminated | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: HISTORY - 1209
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure; Left Bundle Branch Block; Heart Disease
Keywords: Cardiac Resynchronization Therapy; Pacing; His Bundle
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with heart failure and wide QRS: Patients undergoing a cardiac resynchronization therapy procedure
  Interventions: Device: Cardiac Pacing

INTERVENTIONS:
Device: Cardiac Pacing

SUMMARY:
The purpose of this acute study is to perform a preliminary investigation of high septal right ventricular pacing in the vicinity of the His bundle region as an alternate or adjunctive means for cardiac resynchronization in patients with heart failure and wide QRS.

DETAILED DESCRIPTION:
The HISTORY Study is an acute, cross-sectional, multi-center, feasibility study with a randomized within patient test sequence designed to characterize the effects of high septal right ventricular pacing in the vicinity of the His bundle region compared to conventional biventricular pacing for cardiac resynchronization therapy.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older
* Patients willing and capable of providing informed consent, participating in all testing associated with this clinical investigation
* Patients undergoing a CRT implant procedure (pacemaker or defibrillator) for one of the following reasons

  * Indicated for a new device
  * Device upgrade
  * Device replacement
  * Lead revision
* Note: recognized indications for CRT-P and CRT-D as of October 2009 are valid for inclusion in this study. Should new indications become approved during the study conduct; those will also be applied within the inclusion criteria.

Exclusion Criteria:

* Patients unwilling or incapable of signing the informed consent, or patients having previously withdrawn their consent
* Patients in AF that cannot be cardioverted for the study
* RBBB pattern
* Sustained, uncontrolled ventricular tachycardia
* Sinus rhythm < 30 bpm or >100 bpm
* Complete AV node block
* Second degree AV block
* Women who are pregnant or plan to become pregnant during the study (method of assessment upon physician's discretion);
* History of (hemorrhagic) cerebro-vascular accident or TIA

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with wide QRS and undergoing a CRT procedure
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong